CLINICAL TRIAL: NCT06105970
Title: Chinese Community Sample of Hierarchical Model of Psychopathology : Validation and Analysis of Underline Trans-diagnostic Risk Factors
Brief Title: Chinese Community Sample of Hierarchical Model of Psychopathology
Status: Recruiting | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Zhen Wang, vice-president, Shanghai Mental Health Center
Other Study IDs: HiTOP001
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Mental Health Issue; Adverse Childhood Experience
Keywords: Hierarchical Model of Psychopathology

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Community sample: Using social media to randomly inviting participants across all regions of China.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — cross sectional study#no intervention

SUMMARY:
By validating Hierarchy Model of psychopathology(HiTOP) in Chinese community samples, this study aims for illumating the problem of diagnostic heterogeneity and high comorbidity within existing psychiatric classification systems in Chinese culture. Concurrently, this study also focuses on exploring trans-diagonostic risk and proctective factors underline HiTOP dimensions.

the main questions it aims to answer are:

1. Explore HiTOP model cultural differences between western culture and eastern culture.
2. Understand the impact of different dimension of adverse childhood experience on HiTOP structure.
3. Investigate the relationship between individual unique psychological variables and psychopathological dimensions.

Participants will receive a detailed survey trying to measure their psychopathology symptoms, adverse childhood experience and psychological variables. This study expects to fallow up participants for 4 years to monitor the symptom changes.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese citizens
2. Years of education > =9 years.
3. age >= 18 years old.

Exclusion Criteria:

(1)Subjects who have insufficient self-awareness, and are unable to obtain complete informed consent, such as: schizophrenia, manic episode of bipolar disorder, severe depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study aims to recruits partcipants across the whole regions of China, with the aim of collecting representative Chinese community sample.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Chinese version of Hierarchy Model of psychopathology | 1 year
  Constructing the Chinese version of Hierarchy Model of psychopathology. Comparing the differences between Chinese version and western version.
Mapping different dimension of adverse childhood experience on Hierarchy Model of psychopathology structure | 1 year

SECONDARY OUTCOMES:
Investigate the relationship between individual unique psychological variables and psychopathological dimensions. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, PhD, MD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, China